CLINICAL TRIAL: NCT03078738
Title: A First-in-Human Randomized, Double-blind, Placebo-controlled, Fed-fasted, Gender, Single and Multiple Ascending Oral Dose Study, to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of OMT-28 in Healthy Subjects
Brief Title: Safety and Pharmacokinetic Study of OMT-28 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Omeicos Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: OMT28-C0101
Record Dates: First submitted 2017-02-16; First posted 2017-03-13 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers
Keywords: OMT-28; Atrial Fibrillation; SAD; MAD; First-in-Man; Cardiovascular
MeSH Terms: conditions — Atrial Fibrillation | interventions — 17,18-epoxy-5,8,11,14-eicosatetraenoic acid; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: SAD, MAD and Gender parts: double blind randomized. Food Effect part: open label, crossover design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- OMT-28-SAD (Experimental): OMT-28-SAD, Single ascending dose levels 1 - 3 of OMT-28 (15, 30, 60 mg) Oral, healthy young male
  Interventions: Drug: OMT-28
- OMT-28-MAD (Experimental): Multiple ascending dose of dose levels 1 - 3 of OMT-28 over 14 days (4, 12, 36 mg) Oral, healthy young male
  Interventions: Drug: OMT-28
- OMT-28- Food Effect (Experimental): Single dose of OMT-28 (4 mg) Oral, healthy young male
  Interventions: Drug: OMT-28
- OMT-28-Gender (Experimental): Single dose of OMT-28 (4 mg) Oral, healthy non-child bearing potential female
  Interventions: Drug: OMT-28
- Placebo-SAD (Placebo Comparator): Single dose levels 1 - 3 of matching placebo, Oral, healthy young male
  Interventions: Other: Matching Placebo
- Placebo MAD (Placebo Comparator): Multiple dose levels 1 - 3 of matching placebo over 14 days Oral, healthy young male
  Interventions: Other: Matching Placebo
- Placebo-Gender (Placebo Comparator): Single dose of matching Placebo Oral, healthy non-child bearing potential female
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: OMT-28 — OMT-28 is a fully synthetic small molecule that belongs to the family of 17,18-epoxyeicosatetraenoic acids (17,18-EEQ) analogs, a natural metabolite of the omega-3 fatty acid eicosapentaenoic acid (EPA).
  Other Names: 17,18-epoxyeicosatetraenoic acid analog
  Arms: OMT-28- Food Effect; OMT-28-Gender; OMT-28-MAD; OMT-28-SAD
Other: Matching Placebo — Microcrystalline cellulose
  Other Names: Microcrystalline cellulose
  Arms: Placebo MAD; Placebo-Gender; Placebo-SAD

SUMMARY:
The aim of this first-in-human study is to assess the safety, tolerability, PK and exploratory pharmacodynamics (PD) of single and multiple oral ascending doses of OMT-28 in healthy male subjects to support further clinical development of OMT-28 in the indication of atrial fibrillation (AF) and to obtain data on food and gender effects of OMT-28 to guide dosing for Phase II trials.

DETAILED DESCRIPTION:
This first-in-human study will be carried out in one study center involving multiple steps. Up to 100 healthy male and female subjects will be enrolled. The study consists of 4 parts:

1. a single ascending dose (SAD) part
2. a multiple ascending dose (MAD) part
3. a single dose, double cross-over food effect (FE) part.
4. a single dose gender effect part (female subjects group) The safety and PK data will be evaluated by the DSMC after each cohort to decide on further dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. In general good physical health as determined by medical and surgical history, physical examination, 12 lead ECG, vital signs, and clinical laboratory tests
2. Normal blood pressure (Systolic Blood Pressure (SBP) between 100 to 140 mmHg (both inclusive); Diastolic Blood Pressure (DBP) ≥55, ≤89 mmHg) measured after 5 min rest in supine position.
3. SAD, MAD, and FE part: male of 18 to 45 years (inclusive) of age.
4. Gender effect part: female of 18 to 45 years (inclusive) of age.

Exclusion Criteria:

1. More than moderate smoker (> 10 cigarettes/day).
2. More than moderate alcohol consumption (> 35 g of ethanol regularly per day or > 245 g regularly per week).
3. Use of any medication
4. One or more key safety laboratory parameters out of normal range Gender effect part Pregnant or breastfeeding women and of childbearing potential Previous assignment to treatment during this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Safety assessed by frequency and nature of treatment-emergent adverse events | From Day 1 to Day 21

SECONDARY OUTCOMES:
Pharmacokinetics (PK) measured by AUC0-t of OMT-28 in plasma in the SAD | From Day 1 to Day 21
Pharmacokinetics (PK) measured by AUC0-∞ of OMT-28 in plasma in the SAD | From Day 1 to Day 21
Pharmacokinetics (PK) measured by Cmax of OMT-28 in plasma in the SAD | From Day 1 to Day 21
Pharmacokinetics (PK) measured by AUC0-24h of OMT-28 in plasma after single dosing in the SAD | From Day 1 to Day 28
Pharmacokinetics (PK) measured by AUC0-τ after multiple dosing on Day 7 and 14 in the MAD | From Day 7 to Day 14
Pharmacokinetics (PK) of OMT28 measured Cmax after multiple dosing on Day 7 and 14 in the MAD | From Day 7 to Day 14
Pharmacokinetics (PK) in Food Effect and Gender Part measured by AUC0-t of OMT-28 in plasma | From Day 1 to Day 21 (Gender) and Day 28 (F&E)
Pharmacokinetics (PK) in Food Effect and Gender Part measured by AUC0-∞ of OMT-28 in plasma | From Day 1 to Day 21 (Gender) and Day 28 (F&E)
Pharmacokinetics (PK) of OMT28 in Food Effect and Gender Part measured by Cmax of OMT-28 in plasma | From Day 1 to Day 21 (Gender) and Day 28 (F&E)
Change-from-baseline of QTcF (∆QTcF) | From baseline to Day 28
Change from-baseline of heart rate | From baseline to Day 28
Change from-baseline of PR interval in ECG | From baseline to Day 28
Change from-baseline of QRS interval (∆HR, ∆PR and ∆QRS) | From baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Frank Schaumann, Dr. med, Principal Investigator — CRS-Mönchengladbach
Locations (1):
- CRS-Mönchengladbach, Mönchengladbach, Germany

IPD SHARING:
Plan to Share IPD: No